CLINICAL TRIAL: NCT00525148
Title: LUX Lung 2 A Phase II Single-arm Trial of BIBW 2992 in Non-small Cell Lung Cancer Patients With EGFR Activating Mutations
Brief Title: LUX Lung 2 Phase II Single Arm BIBW 2992 "Afatinib" in NSCLC With EGFR Activating Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.22
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental): Patients start continuous once daily oral treatment of BIBW 2992 at high dose, until progression or undue Adverse Events (AEs) develop. Patients can be dose-reduced up to two times if needed after temporary discontinuation of treatment due to drug-related AEs. After protocol amendment 2 (17 Dec 2008), the starting dose of BIBW 2992 was reduced to a medium dose, with 2 possible dose reductions if needed after discontinuation due to drug-related AEs.
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — This is an open label study. Patients are treated with BIBW 2992 until disease progression or undue AEs

SUMMARY:
The primary objective of this open-label, single arm Phase II trial is to explore the efficacy of BIBW 2992 defined by the objective response rate (CR, PR) as determined by RECIST criteria in patients with advanced NSCLC Stage IIIB or IV whose tumors harbor activating mutations within exon 18 to exon 21 of the EGFR receptor. Patients progressing or relapsing after one prior cytotoxic chemotherapy regimen as well as chemotherapy naïve patients (only in stage 2) will be allowed to enter into the trial.

ELIGIBILITY:
Inclusion criteria:

1. Patients with pathologically confirmed diagnosis of NSCLC Stage IIIB (with pleural effusion) adenocarcinoma or Stage IV adenocarcinoma.
2. Presence of activating mutation(s) in exon 18 to exon 21 of the EGFR-receptor confirmed by direct DNA sequencing of NSCLC tumor tissue.
3. Progressive disease following a first line cytotoxic chemotherapy regimen or have recurrent disease after prior neoadjuvant or adjuvant chemotherapy. Patients who have not received first-line cytotoxic chemotherapy can be enrolled in stage 2 of the trial, if the criteria for entering stage 2 are met.
4. Patients with at least one tumor lesion that can accurately be measured by computed tomography (CT) or magnetic resonance imaging (MRI) in at least one dimension with longest diameter to be recorded as 20 mm using conventional techniques or 10 mm with spiral CT scan.
5. Male or female patient aged 18 years.
6. Life expectancy of at least three (3) months.
7. Written informed consents that is consistent with ICH-GCP guidelines.
8. Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2.

Exclusion criteria:

1. More than one (1) prior cytotoxic chemotherapy treatment regimen for relapsed or metastatic NSCLC.
2. Chemo-, hormone- (other than Megace®) or immunotherapy within the past 4 weeks or within less than four half-lives of the previous drug prior to treatment with the trial drug and/or persistence of toxicities of prior anticancer therapies which are deemed to be clinically relevant.
3. Previous treatment with erlotinib (Tarceva®), gefitinib (Iressa®) or any other EGFR inhibiting small molecule or antibody.
4. Brain metastases, which are symptomatic; patients with treated, asymptomatic brain metastases are eligible with stable brain disease for at least four (4) weeks without the requirement for steroids or anti-epileptic therapy.
5. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohns disease, malabsorption, or CTCAE Grade >2 diarrhea of any etiology at baseline.
6. Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
7. Other malignancies diagnosed within the past five (5) years (other than non-melanomatous skin cancer and in situ cervical cancer).
8. Radiotherapy within the past 2 weeks prior to treatment with the trial drug.
9. Patients with any serious active infection (i.e., requiring an IV antibiotic, antifungal, or antiviral agents).
10. Patients with known HIV, active hepatitis B or active hepatitis C.
11. Known or suspected active drug or alcohol abuse.
12. Women of child-bearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial.
13. Pregnancy or breast feeding.
14. Patient unable to comply with the protocol.
15. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3.
16. Cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram.
17. QTc interval greater than 0.47 second.
18. Prior treatment with anthracyclines with a cumulative dose of doxorubicin (or equivalent) greater than 400 mg/m2.
19. Absolute neutrophil count (ANC) less than 1500/mm3.
20. Platelet count less than 100 000 /mm3.
21. Bilirubin greater than 1.5 mg / dl (greater than 26 micromol / L, SI unit equivalent).
22. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal).
23. Serum creatinine greater than 1.5 times of the upper normal limit or calculated/measured creatinine clearance equal or less than 45 ml / min.
24. Patients with known pre-existing interstitial lung disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- United States (23):
  - 1200.22.28 Boehringer Ingelheim Investigational Site, Bakersfield, California
  - 1200.22.32 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1200.22.4 Boehringer Ingelheim Investigational Site, Mission Hills, California
  - 1200.22.16 Boehringer Ingelheim Investigational Site, Orange, California
  - 1200.22.19 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1200.22.29 Boehringer Ingelheim Investigational Site, North Miami Beach, Florida
  - 1200.22.10 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1200.22.18 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1200.22.3 Boehringer Ingelheim Investigational Site, Bethesda, Maryland
  - 1200.22.14 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.22.24 Boehringer Ingelheim Investigational Site, Flint, Michigan
  - 1200.22.5 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1200.22.15 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.22.26 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.22.1 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1200.22.27 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 1200.22.25 Boehringer Ingelheim Investigational Site, Valhalla, New York
  - 1200.22.6 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1200.22.7 Boehringer Ingelheim Investigational Site, Wynnewood, Pennsylvania
  - 1200.22.22 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1200.22.31 Boehringer Ingelheim Investigational Site, Fairfax, Virginia
  - 1200.22.40 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 1200.22.33 Boehringer Ingelheim Investigational Site, Seattle, Washington
- Taiwan (7):
  - 1200.22.88604 Taichung Veterans General Hospital, Taichung
  - 1200.22.88605 China Medical University Hospital, Taichung
  - 1200.22.88606 Boehringer Ingelheim Investigational Site, Tainan
  - 1200.22.88601 National Taiwan University Hospital, Taipei
  - 1200.22.88602 Veterans General Hospital, Taipei
  - 1200.22.88607 Boehringer Ingelheim Investigational Site, Taipei
  - 1200.22.88603 Chang Gung Memorial Hosp-Linkou, Taoyuan District

REFERENCES:
- [Derived] Yang JC, Sequist LV, Geater SL, Tsai CM, Mok TS, Schuler M, Yamamoto N, Yu CJ, Ou SH, Zhou C, Massey D, Zazulina V, Wu YL. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2, LUX-Lung 3, and LUX-Lung 6. Lancet Oncol. 2015 Jul;16(7):830-8. doi: 10.1016/S1470-2045(15)00026-1. Epub 2015 Jun 4. PMID 26051236
- [Derived] Yang JC, Shih JY, Su WC, Hsia TC, Tsai CM, Ou SH, Yu CJ, Chang GC, Ho CL, Sequist LV, Dudek AZ, Shahidi M, Cong XJ, Lorence RM, Yang PC, Miller VA. Afatinib for patients with lung adenocarcinoma and epidermal growth factor receptor mutations (LUX-Lung 2): a phase 2 trial. Lancet Oncol. 2012 May;13(5):539-48. doi: 10.1016/S1470-2045(12)70086-4. Epub 2012 Mar 26. PMID 22452895

RESULTS

PARTICIPANT FLOW:
Groups:
- First-line Afatinib 40 mg: First-line patients were enrolled after Amendment 1 with a starting oral dose of Afatinib 40 mg daily after Amendment 2. Dose reduction scheme was defined for patients unable to tolerate this dose.
- First-line Afatinib 50 mg: First-line patients were enrolled after Amendment 1 with a starting oral dose of Afatinib 50 mg daily. Dose reduction scheme was defined for patients unable to tolerate this dose.
- Second-line Afatinib 40 mg: Second-line patients received a starting oral dose of Afatinib 40 mg daily only after Amendment 2. Dose reduction scheme was defined for patients unable to tolerate this dose.
- Second-line Afatinib 50 mg: Second-line patients received a starting oral dose of Afatinib 50 mg daily. Dose reduction scheme was defined for patients unable to tolerate this dose.
Period: Overall Study
Arm/Group | First-line Afatinib 40 mg | First-line Afatinib 50 mg | Second-line Afatinib 40 mg | Second-line Afatinib 50 mg
Started | 23 (entered and treated) | 38 (entered and treated) | 7 (entered and treated) | 61 (entered and treated)
Completed | 0 | 0 | 0 | 0
Not Completed | 23 | 38 | 7 | 61
Not completed — Other Adverse Event | 3 | 5 | 1 | 8
Not completed — Progressive disease | 18 | 30 | 6 | 49
Not completed — Refused continuation of study medication | 0 | 2 | 0 | 1
Not completed — Other than stated | 2 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Treated set: The patients who had taken at least one dose of afatinib were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | First-line Afatinib 40 mg | First-line Afatinib 50 mg | Second-line Afatinib 40 mg | Second-line Afatinib 50 mg | Total
Number analyzed (Participants) | 23 | 38 | 7 | 61 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.0) | 62 (9.6) | 57 (14.5) | 61 (11.5) | 62 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 27 | 3 | 32 | 75
  Male | 10 | 11 | 4 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) as Determined by RECIST 1.0
Description: Objective response (OR) was assessed for all treated patients by independent review as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. OR included complete response (CR) and partial response (PR), where CR or PR must have been confirmed by a subsequent response in ≥28 days.
Time Frame: Response assessment is done at end of Week 4 (after Course 1), Week 8 (after Course 2), Week 12 (after Course 3) and at 8-week intervals thereafter, up to 93 months.
Population: Treated set: The patients who had taken at least one dose of afatinib were included in the treated set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Afatinib: Patients in the four initial cohorts are combined in the efficacy presentations. Patients start once daily oral treatment of BIBW 2992 (Afatinib) at 50 mg before protocol amendment 2 (17 Dec 2008), until progression or undue adverse events (AEs) development. Patients can be dose-reduced up to two times if needed after temporary interruption of treatment due to drug- related AEs. After protocol amendment 2, the starting dose of BIBW 2992 was reduced to 40 mg, with 2 possible dose reductions if needed after temporary dose interruption due to drug-related AEs.
Arm/Group | Afatinib
Number analyzed (Participants) | 129
percentage of participants | 62.0 [53.1 to 70.4]

2. Secondary Outcome: Clinical Benefit as Determined by RECIST 1.0
Description: Clinical benefit was evaluated according to RECIST 1.0 by independent review assessment. Patients whose best RECIST 1.0 assessment was stable disease (SD), partial response (PR), or complete response (CR) were considered to have derived a clinical benefit from treatment.
Time Frame: as for outcome 1
Population: Treated set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 129
Percentage of participants | 82.2 [74.5 to 88.3]

3. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit (disease control) as per independent review was defined as the time from the start of treatment to the time of progression or death (whichever occurred first), among patients with evidence of SD, PR or CR.
Time Frame: as for outcome 1
Population: Treated Set
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Afatinib
Number analyzed (Participants) | 129
weeks | 81.6 (80.5) [74.5 to 88.3]

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response (OR) was measured from the time the criteria for CR or PR (whichever was documented first) were first met until the first date that progressive disease or death (or date of censoring for PFS) was objectively documented as per independent review.
Time Frame: as for outcome 1
Population: Treated set including only patients with objective response.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib
Number analyzed (Participants) | 80
Weeks | 76.5 (77.2)

5. Secondary Outcome: Time to Objective Response
Description: Time to objective response was defined as the number of days from the start of treatment to the first recorded objective response. Patients who did not experience objective response during the study were censored at the time of treatment discontinuation.
  The results are provided as the percentage of participants for this Outcome Measure.
Time Frame: as for outcome 1
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 129
Percentage of participants
  Week 4 | 38.8
  Week 8 | 12.4
  Week 12 | 1.6
  Week 20 | 5.4
  Week 28 | 0.0
  Week 36 | 1.6
  Week 44 | 0.0
  >= Week 52 | 2.3
  no objective response | 38.0

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) as per independent review was defined as the duration of time from the start of treatment until the day of objective tumor progression was confirmed by tumor imaging (Progressive Disease according to RECIST 1.0) or death, whichever came first. Patients with unknown progression status or unknown date of progression were reviewed on a case-by-case basis. Patients known to be alive without progression at the end of the trial or the last follow-up visit were censored at the date of the last imaging when the patient was known to be alive and progression-free. Medians are calculated from the Kaplan-Meier estimates and 95% confidence intervals, using Greenwood's standard error estimate.
Time Frame: as for outcome 1
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib
Number analyzed (Participants) | 129
Months | 10.2 [8.1 to 13.7]

7. Secondary Outcome: Overall Survival Time
Description: Overall survival time (OS) was also evaluated and was defined as the duration of time from start of treatment to time of death up to 93 months, regardless of the cause of death. Medians are calculated from the Kaplan-Meier estimates and 95% confidence intervals, using Greenwood's standard error estimate.
Time Frame: Start of treatment to time to all death, up to 93 months
Population: Treated set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib
Number analyzed (Participants) | 129
Months | 26.8 [22.0 to 34.5]

8. Secondary Outcome: Cpre,ss,29
Description: Predose concentration of the analyte in plasma at steady state immediately before administration of the 29th dose (Cpre,ss,29).
Time Frame: -0:05h (pre-dose) on Day 29
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 30 mg: Subjects receiving 30 mg of Afatinib daily.
- Afatinib 40 mg: Subjects receiving 40 mg of Afatinib daily.
- Afatinib 50 mg: Subjects receiving 50 mg of Afatinib daily.
Arm/Group | Afatinib 30 mg | Afatinib 40 mg | Afatinib 50 mg
Number analyzed (Participants) | 3 | 38 | 60
ng/mL | 54.1 (78.5) | 27.9 (63.1) | 33.7 (64.1)

9. Secondary Outcome: Safety of BIBW 2992 as Indicated by Incidence of Specified Adverse Events.
Description: Safety of afatinib as indicated by incidence of specified adverse events: skin reactions (a preferred term of the system organ class: Skin and subcutaneous tissue disorders) and gastrointestinal (GI) (a system organ class).
Time Frame: First administration of trial medication until 28 days after last administration of trial medication, up to 93 months.
Population: Treated set
Measure: Number; unit: Percentage of participants
Groups:
- BIBW 40mg: Subjects receiving starting doses 40 mg of Afatinib daily.
- BIBW 50mg: Subjects receiving starting doses 50 mg of Afatinib daily.
Arm/Group | BIBW 40mg | BIBW 50mg
Number analyzed (Participants) | 30 | 99
Percentage of participants
  skin reactions | 16.7 | 27.3
  gastrointestinal (GI) | 100.0 | 97.0

10. Secondary Outcome: Safety of BIBW 2992 as Indicated by Intensity and Incidence of Worst Adverse Events Graded According to NCI CTCAE Version 3.0
Description: Safety of afatinib as indicated by intensity and incidence of worst adverse events graded according to National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) Version 3.0 (R04-0474).
Time Frame: First administration of trial medication until 28 days after last administration of trial medication, up to 93 months.
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | BIBW 40mg | BIBW 50mg
Number analyzed (Participants) | 30 | 99
Percentage of participants
  Grade 1 | 3.3 | 1.0
  Grade 2 | 36.7 | 25.3
  Grade 3 | 46.7 | 57.6
  Grade 4 | 6.7 | 3.0
  Grade 5 | 6.7 | 12.1

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication, up to 93 months.
Arm/Group | BIBW 40mg | BIBW 50mg
Serious Adverse Events (participants affected / at risk) | 9/30 | 44/99
Other Adverse Events (participants affected / at risk) | 30/30 | 98/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBW 40mg (N=30) | BIBW 50mg (N=99)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cyst rupture (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Pneumonia bacterial (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Biopsy prostate normal (Investigations) | 0 | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 4
Seizure (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBW 40mg (N=30) | BIBW 50mg (N=99)
Anaemia (Blood and lymphatic system disorders) | 1 | 10
Blepharitis (Eye disorders) | 2 | 2
Dry eye (Eye disorders) | 2 | 5
Eye pruritus (Eye disorders) | 2 | 1
Vision blurred (Eye disorders) | 0 | 9
Abdominal distension (Gastrointestinal disorders) | 2 | 10
Abdominal pain upper (Gastrointestinal disorders) | 2 | 17
Cheilitis (Gastrointestinal disorders) | 2 | 11
Constipation (Gastrointestinal disorders) | 3 | 21
Diarrhoea (Gastrointestinal disorders) | 29 | 92
Dry mouth (Gastrointestinal disorders) | 0 | 11
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Eructation (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 7
Haematochezia (Gastrointestinal disorders) | 0 | 5
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 5
Haemorrhoids (Gastrointestinal disorders) | 0 | 8
Melaena (Gastrointestinal disorders) | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 4 | 35
Nausea (Gastrointestinal disorders) | 4 | 16
Oral pain (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 37
Vomiting (Gastrointestinal disorders) | 8 | 16
Asthenia (General disorders) | 4 | 5
Chest pain (General disorders) | 2 | 8
Fatigue (General disorders) | 8 | 25
Mucosal inflammation (General disorders) | 8 | 39
Oedema peripheral (General disorders) | 7 | 11
Pain (General disorders) | 2 | 5
Pyrexia (General disorders) | 2 | 11
Xerosis (General disorders) | 4 | 2
Cellulitis (Infections and infestations) | 0 | 7
Conjunctivitis (Infections and infestations) | 2 | 23
Folliculitis (Infections and infestations) | 7 | 36
Herpes virus infection (Infections and infestations) | 2 | 1
Oral candidiasis (Infections and infestations) | 2 | 3
Paronychia (Infections and infestations) | 20 | 79
Pyuria (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 3
Tinea pedis (Infections and infestations) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 19
Urinary tract infection (Infections and infestations) | 5 | 17
Alanine aminotransferase increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 7
Weight decreased (Investigations) | 3 | 19
Decreased appetite (Metabolism and nutrition disorders) | 10 | 39
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 9
Dizziness (Nervous system disorders) | 10 | 20
Dysgeusia (Nervous system disorders) | 2 | 10
Headache (Nervous system disorders) | 6 | 16
Hypoaesthesia (Nervous system disorders) | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 3 | 25
Dysuria (Renal and urinary disorders) | 0 | 6
Haematuria (Renal and urinary disorders) | 1 | 5
Pollakiuria (Renal and urinary disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 41
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 26
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 22
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 46
Acne (Skin and subcutaneous tissue disorders) | 7 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 15
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 35
Eczema (Skin and subcutaneous tissue disorders) | 3 | 9
Erythema (Skin and subcutaneous tissue disorders) | 0 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 8
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 60
Rash (Skin and subcutaneous tissue disorders) | 20 | 75
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 10
Skin fissures (Skin and subcutaneous tissue disorders) | 8 | 26
Skin reaction (Skin and subcutaneous tissue disorders) | 5 | 27
Haemorrhage (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.